CLINICAL TRIAL: NCT04368052
Title: Evaluation of The Association Between Cognitive Dysfunction and Brain Cellular Damage During Liver Transplantations
Brief Title: Liver Transplant Does it Affect the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mustafa Nuri Deniz, Assoc. Prof, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 27042020
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Brain Damage; Postoperative Cognitive Dysfunction; Neuron Specific Enolase; Glial Fibrillary Acidic Protein
Keywords: Liver transplantation; Neuronal damage; Brain; Biochemical marker; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Brain Injuries; Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation (Other): preoperative and postoperative cognitive functions of 33 patients undergoing liver transplantation (LTx) were measured using the Mini Mental Test (MMT) whereas simultaneous neuronal damage was evaluated through the measurement of S-100 beta (S100β), Neuron specific enolase (NSE) and Glial fibrillary acidic protein (GFAP) levels.
  Interventions: Diagnostic Test: Mini Mental Test (MMT), S-100 beta, Neuron specific enolase and Glial fibrillary acidic protein

INTERVENTIONS:
Diagnostic Test: Mini Mental Test (MMT), S-100 beta, Neuron specific enolase and Glial fibrillary acidic protein — Patients undergoing liver transplantation (LTx) were measured using the Mini Mental Test (MMT) whereas simultaneous neuronal damage was evaluated through the measurement of S-100 beta (S100β), Neuron specific enolase (NSE) and Glial fibrillary acidic protein (GFAP) levels.

SUMMARY:
Neuronal damage caused by neuroinflammation in patients undergoing major surgery is the most determinant factor of postoperative cognitive disfunction (POCD). Neuronal damage can be detected through the measurement of biochemical markers of brain damage. The aim of this study was to evaluate neuronal damage and its association with POCD during liver transplantations. After the approval of the ethics committee and patient consents, preoperative and postoperative cognitive functions of 33 patients undergoing liver transplantation (LTx) were measured using the Mini Mental Test (MMT) whereas simultaneous neuronal damage was evaluated through the measurement of S-100 beta (S100β), Neuron specific enolase (NSE) and Glial fibrillary acidic protein (GFAP) levels. As a result, there was no statistically significant difference between preoperative and postoperative MMTs. However, there was a statistically significant decrease in postoperative GFAP and a statistically significant increase in NSE compared to preoperative values. The decrease in S100β level was statistically insignificant. In conclusion, neuroprotective approaches in the investigator's anesthesia protocol protect patients from brain damage during liver transplantation and prevent the development of POCD, which was indicated by the insignificant change in MMT scores and S100β level and the significant decrease in GFAP. Since the significant increase in NSE levels during liver transplantations was deemed to might have been associated with causes other than neuronal damage, NSE should not be evaluated as a marker of brain damage in these operations.

ELIGIBILITY:
Inclusion Criteria:

* Score of 23 or above on the Mini Mental Test (MMT) conducted in the preparation room prior to the operation,
* No gastrointestinal bleeding in the last 1 month
* No history of neuroactive drug use
* Consented for the study.

Exclusion Criteria:

* Hepatic encephalopathy,
* Neurological disorder
* Psychiatric disorder,

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Neuron specific enolase (NSE) | Throughout the operation
  NSE should not be evaluated as a marker of brain damage in liver transplantations.

SECONDARY OUTCOMES:
S-100 beta (S100β), and Glial fibrillary acidic protein (GFAP) | Throughout the operation
  Neuroprotective approach protects patients from brain damage during liver transplantation and prevent the development of POCD, which was indicated by the insignificant change in MMT scores and S100β level and the significant decrease in GFAP.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Sezer, Assoc. Prof., Principal Investigator — Ege University Medical Faculty, Department of Medical Biochemistry
Locations (1):
- Ege University Faculty of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No